CLINICAL TRIAL: NCT03934606
Title: Evaluating an Alternative Clinical Genetics Cancer Care Deliver Model: A Pilot Study of Patient Outcomes
Brief Title: Evaluating an Alternative Clinical Genetics Cancer Care Deliver Model
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 15917; 828314 (Other: IRB)
Record Dates: First submitted 2019-02-13; First posted 2019-05-02 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Pancreas Cancer; Prostate Cancer; Hereditary Cancer; Genetic Predisposition to Disease
MeSH Terms: conditions — Pancreatic Neoplasms; Prostatic Neoplasms; Genetic Predisposition to Disease | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Genetic testing for hereditary predisposition — Change in distress levels (HADS-Anxiety) from Baseline to Assessments #2 and #3, measured as an effect size among participants who receive a pathogenic variant(s), no pathogenic variant(s), and variant(s) of uncertain significance
  Other Names: Behavioral Assessments

SUMMARY:
To evaluate an alternative clinical genetics cancer care delivery model, using non-genetic providers to introduce and order genetic testing. 250 prostate and 250 pancreatic patients will be recruiting. They will undergo genetic testing and complete study questionnaires. Results from this pilot study will be used to inform the strategies used by the Clinical Risk Evaluation Program (CREP) Genetic Counelors (CGS) and GI/GU physicians to deliver genetic testing and return genetic risk information to patients with prostate or pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* • Penn patient age 18 years or older.

  * Diagnosed with prostate cancer or pancreas cancer.
  * Deemed to be clinically appropriate for multiplex genetic testing by their Urologic Cancer Program (GU) physician or Gastrointestinal Cancer Program (GI) physician at the Abramson Cancer
  * Agreed to receive clinical multiplex genetic testing from their physician.
  * English-fluent; the surveys were designed and validated in English and are not currently available in other languages.

Exclusion Criteria:

* • Patients who do not or will not receive their ongoing cancer care at Penn

  * Major psychiatric illness or cognitive impairment that in the judgment of the study investigators or study staff would preclude study participation.
  * Any patients who are unable to comply with the study procedures as determined by the study investigators or study staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen at Penn Medicine with a pancreas cancer or metastatic prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1488 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
baseline to post-results change in distress levels | 1-3months
  Change in distress levels (HADS-Anxiety) from Baseline to Time point #2 (post-disclosure) measured as an effect size among participants who receive a pathogenic variant(s), no pathogenic variant(s), and variant(s) of uncertain significance
baseline to post-results change in distress levels | 3 months
  Change in distress levels (HADS-Anxiety) from Baseline to Time point #3 (3 months post-disclosure) measured as an effect size among participants who receive a pathogenic variant(s), no pathogenic variant(s), and variant(s) of uncertain significance

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Medicine - University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided